CLINICAL TRIAL: NCT01186146
Title: Optimal Duration of Clopidogrel Therapy After Drug-Eluting Stent Implantation to Reduce Late Coronary Arterial Thrombotic Events
Brief Title: Duration of Clopidogrel Therapy After Drug-Eluting Stent (DES-LATE)
Acronym: DES-LATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0186
Record Dates: First submitted 2010-08-17; First posted 2010-08-23 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary disease; stents; antiplatelet drugs; drug-eluting stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): Aspirin monotherapy (stopping clopidogrel at 1 year after DES)
  Interventions: Drug: Aspirin monotherapy
- Aspirin,Clopidogrel (Experimental): Aspirin,Clopidogrel Dual antiplatelet therapy (continue aspirin and clopidogrel 1year after DES)
  Interventions: Drug: Aspirin,Clopidogrel

INTERVENTIONS:
Drug: Aspirin monotherapy — stopping clopidogrel at 1 year after DES
  Arms: Aspirin
Drug: Aspirin,Clopidogrel — continue aspirin and clopidogrel 1year after DES
  Other Names: Aspirin,Clopidogrel Dual antiplatelet therapy
  Arms: Aspirin,Clopidogrel

SUMMARY:
This is randomized-controlled trial to evaluate the difference of composite of cardiac death, myocardial infarction, or Stroke between the dual antiplatelet therapy group and the aspirin monotherapy group after 1-year of drug-eluting stents implantation.

DETAILED DESCRIPTION:
This is subsequent clinical trial of previously published pooled analysis of the REAL-LATE and the ZEST-LATE Trial, in which nonsignificant higher trend for increased rate of death (all-cause and cardiac), myocardial infarction, or stroke in the dual antiplatelet therapy group compared to the aspirin monotherapy group was noted.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients had undergone DES implantation at least 12 months before enrollment, had not had a MACE (death, MI, stroke, or repeat revascularization) or major bleeding, and were dual-therapy at the time of enrollment.
* 2. Time for index PCI to randomization: 12-18 months

Exclusion Criteria:

* Contraindications to the use of antiplatelet drugs (e.g., a concurrent bleeding diathesis or a history of major bleeding)
* Concomitant vascular disease requiring long-term use of clopidogrel
* Other established indications for clopidogrel therapy (e.g., a recent ACS).
* Noncardiac coexisting conditions with a life expectancy < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The composite of cardiac death, myocardial infarction, or stroke | at 2 year after randomization

SECONDARY OUTCOMES:
death | at 2 year after randomization
myocardial infarction | at 2 year after randomization
stroke | at 2 year after randomization
stent thrombosis | at 2 year after randomization
Thrombolysis In Myocardial Infarction (TIMI) major/minor bleeding | at 2 year after randomization
Target Vessl revascularization | at 2 year after randomization
Target Lesion Revascularization | at 2 year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (19):
- South Korea (19):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Busan Saint Mary's Hospital, Busan
  - Cheongju Saint Mary's Hospital, Cheongju-si
  - Chungju ST.Mary's Hospital, Cheongju-si
  - Kangwon National University Hospital, Chooncheon
  - Daegu Catholic University Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - Chonnam National University Hospital, Gwangju
  - DongGuk University Gyongju Hospital, Gyongju
  - NHIC Ilsan Hospital, Ilsan
  - Chonbuk National University Hospital, Jeonju
  - Asan Medical Center, Seoul
  - Catholic University, Kangnam St. Mary's Hospital, Seoul
  - Hangang Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea Veterans Hospital, Seoul
  - St.Mary's Catholic Medical Center, Seoul

REFERENCES:
- [Derived] Lee CW, Ahn JM, Park DW, Kang SJ, Lee SW, Kim YH, Park SW, Han S, Lee SG, Seong IW, Rha SW, Jeong MH, Lim DS, Yoon JH, Hur SH, Choi YS, Yang JY, Lee NH, Kim HS, Lee BK, Kim KS, Lee SU, Chae JK, Cheong SS, Suh IW, Park HS, Nah DY, Jeon DS, Seung KB, Lee K, Jang JS, Park SJ. Optimal duration of dual antiplatelet therapy after drug-eluting stent implantation: a randomized, controlled trial. Circulation. 2014 Jan 21;129(3):304-12. doi: 10.1161/CIRCULATIONAHA.113.003303. Epub 2013 Oct 4. PMID 24097439